CLINICAL TRIAL: NCT02293239
Title: Effects of Whole-Body Electromyostimulation (WB-EMS) Combined With Individualized Nutritional Support on Patients With Malignant Disease Undergoing Curative or Palliative Anti-cancer Treatment
Brief Title: Effects of WB-EMS and Dietetic Treatment on Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMS Tumor 01
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Cancer Cachexia; Weight Loss; Muscle Loss; Muscle Weakness
Keywords: whole-body electromyostimulation; cachexia; cancer; skeletal muscle mass; nutrition
MeSH Terms: conditions — Neoplasms; Weight Loss; Muscular Atrophy; Muscle Weakness; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): "usual care" control group receives individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight)
- WB-EMS group (Experimental): physical exercise group regular WB-EMS training (2 EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight)
  Interventions: Other: Whole-Body Electromyostimulation (WB-EMS)

INTERVENTIONS:
Other: Whole-Body Electromyostimulation (WB-EMS) — WB-EMS training is performed 2x/week for 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
  Arms: WB-EMS group

SUMMARY:
This study evaluates the effects of a 12-week whole-body electromyostimulation (WB-EMS) training combined with individualized nutritional support on body composition, muscle strength and function and quality of life of patients with malignant disease undergoing curative or palliative anti-cancer treatment

ELIGIBILITY:
Inclusion Criteria:

* malignant disease (solid or hematological cancer): head and neck cancer, colorectal carcinoma, small intestinal cancer, gastric cancer, oesophageal cancer, pancreas carcinoma, liver cell carcinoma, cholangiocarcinoma,lung cancer, breast cancer, cervix cancer, ovarian cancer, prostate cancer, renal cell carcinoma, malignant melanoma, patients with leukaemia and malignant lymphomas or Graft-versus-Host-Disease after bone marrow transplantation
* ongoing or planned curative or palliative anti-cancer therapy

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention trials
* acute cardiovascular events
* use of anabolic medications
* epilepsy
* severe neurological diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass | 12 weeks
  Skeletal muscle mass assessed by bioelectrical impedance analysis (in kg)
Physical function - Gait pattern | 12 weeks
  Sensor-based gait analysis

SECONDARY OUTCOMES:
Physical function - Isometric muscle strength | 12 weeks
  Hand grip strength assessed by hand dynamometer (in kg)
Physical function - Endurance | 12 weeks
  Six-minute-walk test (walking distance in m)
Physical function - Lower limb strength | 12 weeks
  30 second sit-to-stand test (number of sit-to-stand cycles)
Patient-reported performance status | 12 weeks
  ECOG performance status/Karnofsky index
Patient-reported Quality of Life (QoL) | 12 weeks
  EORTC QLQ - C30 questionnaire
Patient-reported Fatigue | 12 weeks
  FACIT-Fatigue scale
Inflammatory blood markers | 12 weeks
  Blood collection and analysis e.g. of C-reactive protein (CRP), Albumin

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Klinik 1, University of Erlangen-Nürnberg, Erlangen, Bavaria / Franconia, Germany

REFERENCES:
- [Derived] Schink K, Reljic D, Herrmann HJ, Meyer J, Mackensen A, Neurath MF, Zopf Y. Whole-Body Electromyostimulation Combined With Individualized Nutritional Support Improves Body Composition in Patients With Hematological Malignancies - A Pilot Study. Front Physiol. 2018 Dec 18;9:1808. doi: 10.3389/fphys.2018.01808. eCollection 2018. PMID 30618820
- [Derived] Schink K, Herrmann HJ, Schwappacher R, Meyer J, Orlemann T, Waldmann E, Wullich B, Kahlmeyer A, Fietkau R, Lubgan D, Beckmann MW, Hack C, Kemmler W, Siebler J, Neurath MF, Zopf Y. Effects of whole-body electromyostimulation combined with individualized nutritional support on body composition in patients with advanced cancer: a controlled pilot trial. BMC Cancer. 2018 Sep 12;18(1):886. doi: 10.1186/s12885-018-4790-y. PMID 30208857